CLINICAL TRIAL: NCT06751095
Title: Effects Of Maitland's Mobilization At Mid Versus End Range On Pain, Range Of Motion And Functional Disability In Patients With Knee Osteoarthritis.
Brief Title: Effects Of Maitland's Mobilization At Mid Versus End Range In Knee Osteoarthritis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0114
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: joint range of motion; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland's Mobilization in End Range (Experimental): End-range mobilization will be performed individually in flexion and extension end range of the tibiofemoral joint(0-135 degree).
  Interventions: Other: Maitland's Mobilization in End range
- Maitland's Mobilization in Mid Range (Experimental): Mid range Maitland's mobilization will be performed in (approx. 50-70° knee flexion) of the tibiofemoral joint.
  Interventions: Other: Maitland's mobilization in Mid range

INTERVENTIONS:
Other: Maitland's Mobilization in End range — End-range mobilization will be performed individually in flexion and extension end range of the tibiofemoral joint .(0-135 degree)
  Arms: Maitland's Mobilization in End Range
Other: Maitland's mobilization in Mid range — Mid range Maitland's mobilization will be performed in (approx. 50-70° knee flexion) of the tibiofemoral joint
  Arms: Maitland's Mobilization in Mid Range

SUMMARY:
Knee Osteoarthritis (OA) is the most common form of arthritis affecting mostly elderly people contributing to major cause of disability worldwide.In knee osteoarthritis Maitland's manual therapy technique could be the most effective technique among all in decreasing pain sensitivity and increasing range of motion in knee OA.The aim of this study to compare effects of Maitland's mobilization at mid range versus end range on pain. range of motion and functional disability in patients with knee OA, providing useful insights for healthcare professionals to optimize treatment strategies and enhance outcomes in this context.

DETAILED DESCRIPTION:
Knee Osteoarthritis (OA) is the most common form of arthritis affecting mostly elderly people contributing to major cause of disability worldwide.In knee osteoarthritis Maitland's manual therapy technique could be the most effective technique among all in decreasing pain sensitivity and increasing range of motion in knee OA.The aim of this study to compare effects of Maitland's mobilization at mid range versus end range on pain. range of motion and functional disability in patients with knee OA, providing useful insights for healthcare professionals to optimize treatment strategies and enhance outcomes in this context.

This Randomized Clinical Trial will be conducted at DHQ Gujrat through consecutive sampling technique on 44 patients which will be allocated using simple random sampling through sealed opaque enveloped into (Group A and Group B).Maitland's mobilization at end range(Group A) incorporates the end range Maitland's mobilization,strengthening exercises, knee isometrics, transcutaneous electrical stimulation(TENS) and heating pad .

Maitland's mobilization in Mid range (Group B) will be treated with Mid range Maitland's mobilization, TENS,strengthening exercises,knee isometrics and heating pad.Outcomes, encompassing pain levels, range of motion(ROM), and functional disability will be evaluated through Visual analogue scale (VAS),Goniometer and WOMAC scale.The treatment plan spans 4 weeks, comprising 3 sessions per week. Data will be analyzed during SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups. Data will be collected at baseline and after 4 weeks of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age between 40 to 60 years.
* Participants of both genders will be included.
* Patient with unilateral/bilateral symptomatic tibiofemoral knee OA.
* Patient suffering from stiffness less than 30 minutes
* Patients with radiologically diagnosed case of grade 2 knee OA according to the Kellgren and Lawrence scale
* Patients with reported peak knee pain of >3 on visual analogue scale (VAS)

Exclusion Criteria:

* Participants with acute inflammation of knee
* Participants with severe degenerative lumbar spine disease e.g spondylolisthesis
* Participants with systemic inflammatory arthritic or neurological conditions
* Participants with intraarticular injection in the prior 3 months
* Participants with unstable heart condition
* Participants with received physical therapy of knee in last 3 months

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 Weeks
  The Numerical Pain Rating Scale (NPRS) is a commonly used self-report measure to assess the intensity of pain experienced by individuals. Participants rate their pain on a numerical scale, typically ranging from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
WOMAC Osteoarthritis INDEX | 4 weeks
  The western Ontario and McMaster Universities Arthritis Index(WOMAC) is widely uses in the evaluation of Hip and Knee Osteoarthritis. It is a self administrated questionnaire consisting of 24 item divided into 3 sub-scales: Pain(5items) ,stiffness(2 items) and physical function (17 items)
Universal Goniometer | 4 weeks
  It will measure range of motion of Knee

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Amjad Dr., DPT, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzuki Y, Iijima H, Tashiro Y, Kajiwara Y, Zeidan H, Shimoura K, Nishida Y, Bito T, Nakai K, Tatsumi M, Yoshimi S, Tsuboyama T, Aoyama T. Home exercise therapy to improve muscle strength and joint flexibility effectively treats pre-radiographic knee OA in community-dwelling elderly: a randomized controlled trial. Clin Rheumatol. 2019 Jan;38(1):133-141. doi: 10.1007/s10067-018-4263-3. Epub 2018 Aug 30. PMID 30167975
- [Background] Steultjens MP, Dekker J, van Baar ME, Oostendorp RA, Bijlsma JW. Range of joint motion and disability in patients with osteoarthritis of the knee or hip. Rheumatology (Oxford). 2000 Sep;39(9):955-61. doi: 10.1093/rheumatology/39.9.955. PMID 10986299
- [Background] Pozsgai M, Udvaracz K, Peter IA, Than P, Nusser N. Effect of single end-range and not end-range Maitland mobilization on pressure pain threshold and functional measures in knee osteoarthritis: randomised, controlled clinical trial. Eur J Phys Rehabil Med. 2022 Oct;58(5):774-783. doi: 10.23736/S1973-9087.22.07506-2. Epub 2022 Sep 12. PMID 36094367